CLINICAL TRIAL: NCT01224106
Title: Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Two Year Study to Evaluate the Effect of Subcutaneous RO4909832 on Cognition and Function in Prodromal Alzheimer's Disease With Option for up to an Additional Two Years of Treatment and an Open-Label Extension With Active Study Treatment
Brief Title: A Study of Gantenerumab in Participants With Prodromal Alzheimer's Disease
Acronym: Scarlet Road
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN25203; 2010-019895-66 (EudraCT Number)
Record Dates: First submitted 2010-10-14; First posted 2010-10-19 (Estimated); Results first posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gantenerumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Parts 1 and 2) (Placebo Comparator): Participants with Alzheimer's disease received Placebo by SC injection every 4 weeks (Q4W) for 104 weeks or approximately 2 years during Part 1 of the study. Participants who completed the Week 104 visit were given an option to continue the treatment received during Part 1, for 2 additional years in Part 2.
  Interventions: Drug: Placebo
- Gantenerumab 105 mg (Parts 1 and 2) (Experimental): Participants with Alzheimer's disease received Gantenerumab 105 mg by SC injection every 4 weeks (Q4W) for 104 weeks or approximately 2 years during Part 1 of the study. Participants who completed the Week 104 visit were given an option to continue the treatment received during Part 1, for 2 additional years in Part 2.
  Interventions: Drug: Gantenerumab
- Gantenerumab 225 mg (Parts 1 and 2) (Experimental): Participants with Alzheimer's disease received Gantenerumab 225 mg by SC injection every 4 weeks (Q4W) for 104 weeks or approximately 2 years during Part 1 of the study. Participants who completed the Week 104 visit were given an option to continue the treatment received during Part 1, for 2 additional years in Part 2.
  Interventions: Drug: Gantenerumab
- Placebo (Parts 1 and 2) switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) (Placebo Comparator): Participants with Alzheimer's disease who had received Placebo by SC injection in Part 1 or Part 2, now received Gantenerumab at doses up to 1200 mg by SC injection every 4 weeks (Q4W) for up to 5 additional years.
  Interventions: Drug: Gantenerumab
- Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE]) (Experimental): Participants with Alzheimer's disease who had received Gantenerumab by SC injection in Part 1 or Part 2, now received Gantenerumab at doses up to 1200 mg by SC injection every 4 weeks (Q4W) for up to 5 additional years.
  Interventions: Drug: Gantenerumab

INTERVENTIONS:
Drug: Gantenerumab — Participants received Gantenerumab at 105 mg , 225 mg, or at doses up to 1200 mg SC injection Q4W.
  Arms: Gantenerumab 105 mg (Parts 1 and 2); Gantenerumab 225 mg (Parts 1 and 2); Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE]); Placebo (Parts 1 and 2) switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE])
Drug: Placebo — Participants received Placebo SC injection Q4W.
  Arms: Placebo (Parts 1 and 2)

SUMMARY:
This multi-center, randomized, double-blind, placebo-controlled parallel-group study will evaluate the effect of gantenerumab (RO4909832) on cognition and functioning and the safety and pharmacokinetics in participants with prodromal Alzheimer's Disease. Participants will be randomized to receive subcutaneous (SC) injections of either gantenerumab or placebo. Participants who consent to be part of the sub study will undergo positron emission tomography (PET) scanning to assess brain amyloid. The anticipated time on study treatment is 104 weeks in Part 1, with an option for an additional up to 2 years of treatment in Part 2, followed by an open-label extension (Part 3) until July 2020.

The dosing for Parts 1 and 2 was stopped after a planned futility interim analysis showed a low probability of meeting the primary outcome measure with the doses studied. The study has converted to open-label to investigate higher gantenerumab doses.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, 50-85 years of age
* Participants with prodromal Alzheimer's disease who are not receiving memantine or cholinesterase inhibitors
* Has a study partner who in the investigator's judgement has frequent and sufficient contact with the participant as to be able to provide accurate information as to the participant's cognitive and functional abilities, who agrees to provide information at clinic visits which require partner input for scale completion
* Has had sufficient education or work experience to exclude mental retardation
* Study partner has noticed a recent gradual decrease in participant's memory (over the last 12 months), which the participant may or may not be aware of
* Screening Mini Mental State Exam (MMSE) score of 24 or above

Additional inclusion criteria for sub study:

* Able and willing to travel to PET imaging center and complete the planned scanning sessions
* Past and planned exposure to ionizing radiation not exceeding safe and permissible levels

Exclusion Criteria:

* Other prior or current neurologic or medical disorder which may currently or during the course of the study impair cognition or psychiatric functioning
* A history of stroke
* A documented history of transient ischemic attack within the last 12 months
* History of schizophrenia, schizoaffective or bipolar disorder
* Currently meets criteria for major depression
* Within the last 2 years, unstable or clinical significant cardiovascular disease (myocardial infarction, angina pectoris)

Additional exclusion criteria for sub study:

* Inclusion in a research and/or medical protocol involving PET ligands or other radioactive agents within 12 months
* Present or planned participation in a research and/or medical protocol involving PET ligands or radioactive agents other than study WN25203
* Have planned or are planning to have exposure to ionizing radiation that in combination with the planned administration with study amyloid PET ligand would result in a cumulative exposure that exceeds local recommended exposure limits

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 799 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (139):
- United States (24):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - University of California, San Diego, La Jolla, California
  - Yale University ADRU, New Haven, Connecticut
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Infinity Clinical Research, Hollywood, Florida
  - Accelerated Enrollment Solutions, Orlando, Florida
  - Roskamp Institute, Inc., Sarasota, Florida
  - Compass Research, The Villages, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Indiana University, Indianapolis, Indiana
  - Boston Center for Memory, Newton, Massachusetts
  - Western Michigan University Homer Stryker M.D. School of Medicine Center for Clinical Research, Kalamazoo, Michigan
  - Neurological Research Center, Hattiesburg, Mississippi
  - Princeton Medical Institute, Princeton, New Jersey
  - Nathan Kline Institute, Orangeburg, New York
  - University of Rochester Medical Center; Monroe Community Hospital, Rochester, New York
  - Alzheimer's Memory Center, Matthews, North Carolina
  - Oregon Health and Science University, Layton Aging and Alzheimer's Disease Center, Portland, Oregon
  - Northeastern Pennsylvania Memory, Plains, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Butler Hospital, Providence, Rhode Island
  - Senior Adults Specialty Research, Austin, Texas
  - Texas Neurology PA, Dallas, Texas
  - Clinical Neuroscience Research Associates, Inc., Bennington, Vermont
- Argentina (9):
  - Hospital Italiano, Buenos Aires
  - IME - Instituto Médico Especializado; Ensayos Clínicos, Buenos Aires
  - ALPI-Inst. de Rehabilitacion Marcelo Fitte, Buenos Aires
  - CEMIC, Buenos Aires
  - Mulieris, CABA
  - Instituto De Neurología Cognitiva - INECO, Caba
  - FLENI, CABA
  - Instituto Kremer, Córdoba
  - CENPIA; Neurología - Psicología, La Plata
- Australia (6):
  - Hornsby Ku-ring-gai Hospital; Division of Rehabilitation & Aged Care, Hornsby, New South Wales
  - Prince of Wales Hospital, Academic Department for Old Age Psychiatry, Randwick, New South Wales
  - Royal Adelaide Hospital; Memory Trials Centre, Adelaide, South Australia
  - The Queen Elizabeth Hospital; Neurology, Woodville, South Australia
  - Heidelberg Repatriation Hospital; Medical and Cognitive Research Centre, Heidelberg West, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- UZ Leuven Gasthuisberg, Leuven, Belgium
- Brazil (5):
  - Hospital das Clinicas - UFPR; Ciencias da Saude, Curitiba, Paraná
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Universidade Federal de Sao Paulo - UNIFESPX; Neurologia, São Paulo, São Paulo
  - Hospital das Clinicas - FMUSP; Psiquiatria, São Paulo, São Paulo
- Canada (7):
  - True North Clinical Research, New Minas, Nova Scotia
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Toronto Memory Program, Toronto, Ontario
  - Centre for Memory and Aging, Toronto, Ontario
  - NeuroSearch Developpements inc, Greenfield Park, Quebec
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Neurological and Psychiatric, Montreal, Quebec
  - CHAUQ - Hôpital Enfant-Jésus, Québec, Quebec
- Chile (2):
  - Biomedica Research Group, Santiago
  - Especialidades Medicas LYS, Santiago
- Czechia (2):
  - St. Anne´s University Hospital; Clinical Trials Department, Brno
  - Vestra Clinics s.r.o., Rychnov nad Kněžnou
- Denmark (2):
  - Aarhus Universitetshospital, Neurologisk Afdeling F, Demensklinikken, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, Koebenhavn Oe
- CRST Oy, Turku, Finland
- France (10):
  - Hopital Avicenne; Neurologie, Bobigny
  - Hopital Pellegrin; Cmrr Aquitaine, Bordeaux
  - Hopital Pierre Wertheimer; Laboratoire De Neuro Psychologie, Bron
  - CHU De Caen; Service De Neurologie Dejerine, Caen
  - Hopital B Roger Salengro; Cmrr Lille, Lille
  - Ch Pitie Salpetriere; Cmrr Ile De France Salpetriere, Paris
  - CHU de Rouen Hopital; Service de Neurologie, Rouen
  - Hop Guillaume Et Rene Laennec; Cmrr St Herblain, Saint-Herblain
  - Hopital Hautepierre; Centre dInvestigation Clinique, Strasbourg
  - Hopital de La Grave, Toulouse
- Germany (11):
  - Univ Berlin; Klin fur Psychi & Psycho Charite, Berlin
  - Universitätsklinikum Bonn; Medizinische Klinik und Poliklinik I; Allgemeine Innere Medizin, Bonn
  - Klinikum Joh.Wolfg.Goethe-UNI Zentrum d. Psychiatrie Klinik f. Psychiatrie Psychosomatik, Frankfurt
  - PANAKEIA - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Zentralinstitut für Seelische Gesundheit Abt.Gerontopsychiatrie, Mannheim
  - Pharmakologisches Studienzentrum, Mittweida
  - Neurologische Praxis Dr. Andrej Pauls, München
  - Klinikum rechts der Isar der TU München; Klinik für Psychiatrie und Psychotherapie, München
  - Office of Dr Klaus Steinwachs Neurology & Psychiatry, Nuremberg
  - Universitätsklinikum Rostock Zentrum für Nervenheilkunde, Rostock
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
- Italy (8):
  - Nuovo Ospedale Civile S. Agostino-Estense; Clinica Neurologica - Dipartimento di Neuroscienze, Modena, Emilia-Romagna
  - Universita' Di Parma Istituto Neurologia, Parma, Emilia-Romagna
  - Azienda Ospedaliera Spedali Civili; Scienze Neurologiche, Brescia, Lombardy
  - IRCCS "Centro S. Giovanni di Dio" Fatebenefratelli -UO Alzheimer, Brescia, Lombardy
  - Irccs Multimedica Santa Maria; Unita' Di Neurologia, Castellanza, Lombardy
  - Fondazione San Raffaele Del Monte Tabor; Dipartimento Di Neurologia, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I-G.M. Lancisi-G. Salesi Di Ancona, Torrette - Ancona, The Marches
  - Uni Di Firenze Dip. Scienze Neurol Psic Sod Neurologia 1, Florence, Tuscany
- Mexico (7):
  - Hospital Mexico Americano, Guadalajara, Mexico CITY (federal District)
  - Hospital Universitario; Dr. Jose E. Gonzalez, Monterrey, Nuevo León
  - Hospital Angeles de Culiacán, Neurociencias Estudios Clínicos SC, Culiacán
  - Unidad de Investigacion en Enfermedades Cronico-Degenerativa; Reumatologia, Guadalajara
  - Estimulacion Magnetica Trnscraneal de Mexico SC., Mexico City
  - Centro Medico San Francisco; Geriatrics, Monterrey
  - Hospital Universitario de Saltillo, Saltillo
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis; Polikliniek Geriatrie, 's-Hertogenbosch
  - Brain Research Center B.V, Amsterdam
- Poland (5):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - PALLMED Sp. z o.o. prowadząca NZOZ DOM SUE RYDER, Bydgoszcz
  - NEURO - KARD Ośrodek Badań Klinicznych, Poznan
  - Przychodnia Specjalistyczna PROSEN, Warsaw
  - mMED Maciej Czarnecki, Warsaw
- Portugal (2):
  - Hospital Prof. Dr. Fernando Fonseca; Servico de Neurologia, Amadora
  - Hospital de Santa Maria; Servico de Neurologia, Lisbon
- Russia (5):
  - State autonomous institution of healthcare Inter-regional clinical and diagnostic center, Kazan'
  - Saint Petersburg State Institution of Healthcare City Geriatric Medico-Social Center, Saint Petersburg
  - Russian Medical Military Academy n.a. S.M.Kirov; Neurology Department, Saint Petersburg
  - City Clinical Hospital # 2 n.a. V.I. Razumovsky, Saratov
  - Sverdlovsk Regional Clinical Psychoneurological War Veteran Hospital, Yekaterinburg
- South Korea (5):
  - Seoul National University Bundang Hospital; Neurology Department, Gyeonggi-do
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Asan Medical Center., Seoul
- Spain (10):
  - Fundació ACE, BArcelon, Barcelona
  - Hospital Mutua De Terrasa; Servicio de Neurologia, Terrassa, Barcelona
  - Hospital de Cruces; Servicio de Neurologia, Barakaldo, Vizcaya
  - Hospital del Mar; Servicio de Neurologia, Barcelona
  - Hospital Clinic i Provincial; Servicio de Neurologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neurologia, Barcelona
  - Hospital Ramon y Cajal; Servicio de Neurologia, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Neurologia, Madrid
  - Hospital Universitario La Paz; Servicio de Neurologia, Madrid
  - Hospital Universitario Dr. Peset; Servicio de Neurologia, Valencia
- Skånes Universitetssjukhus Malmö, Minneskliniken, Malmo, Sweden
- Switzerland (2):
  - Felix Platter-Spital Medizin Geriatrie, Basel
  - HUG; Département de santé mentale et de psychiatrie Unité de psychiatrie gériatrique, Chêne-Bourg
- Turkey (Türkiye) (3):
  - Akdeniz University School of Medicine, Neurology Department, Antalya
  - Istanbul University Istanbul School of Medicine; Neurology, Istanbul
  - Ondokuz Mayis University School of Medicine; Neurology, Samsun
- United Kingdom (9):
  - Addenbrooke's Hospital, Cambridge
  - Llandough Hospital; Llandough Hospital Memory Team 3rd Floor Academic Building, Cardiff
  - St Margaret's Hospital, Epping
  - Glasgow Memory Clinic, Glasgow
  - Charing Cross Hospital; Dept of Neurosciences, London
  - Campus for Ageing & Vitality; Clincal Ageing Research Unit, Newcastle
  - Moorgreen Hospital; Memory Assessment & Rsch Ctr, Southampton
  - Victoria Centre; Kingshill Research Centre, Swindon
  - Hollins Park Hospital, Warrington

REFERENCES:
- [Derived] Boada M, Neve A, Das B, Wojtowicz J, Huang Z, Bullain S, Watkin M, Lott D, Bittner T, Delmar P, Klein G, Hofmann C, Kerchner GA, Smith J, Baudler M, Fontoura P, Doody RS. Long-term safety of gantenerumab in participants with Alzheimer's disease: A phase III, open-label extension study (SCarlet RoAD). J Alzheimers Dis. 2025 Jan;103(2):528-541. doi: 10.1177/13872877241303644. Epub 2024 Dec 16. PMID 39686620
- [Derived] Klein G, Delmar P, Voyle N, Rehal S, Hofmann C, Abi-Saab D, Andjelkovic M, Ristic S, Wang G, Bateman R, Kerchner GA, Baudler M, Fontoura P, Doody R. Gantenerumab reduces amyloid-beta plaques in patients with prodromal to moderate Alzheimer's disease: a PET substudy interim analysis. Alzheimers Res Ther. 2019 Dec 12;11(1):101. doi: 10.1186/s13195-019-0559-z. PMID 31831056
- [Derived] Ostrowitzki S, Lasser RA, Dorflinger E, Scheltens P, Barkhof F, Nikolcheva T, Ashford E, Retout S, Hofmann C, Delmar P, Klein G, Andjelkovic M, Dubois B, Boada M, Blennow K, Santarelli L, Fontoura P; SCarlet RoAD Investigators. A phase III randomized trial of gantenerumab in prodromal Alzheimer's disease. Alzheimers Res Ther. 2017 Dec 8;9(1):95. doi: 10.1186/s13195-017-0318-y. PMID 29221491
- [Derived] Delrieu J, Ousset PJ, Vellas B. Gantenerumab for the treatment of Alzheimer's disease. Expert Opin Biol Ther. 2012 Aug;12(8):1077-86. doi: 10.1517/14712598.2012.688022. Epub 2012 May 15. PMID 22583155 (Retraction: PMID 34856846 Expert Opin Biol Ther. 2021 Dec;21(12):1-2)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 128 centers in 24 countries.
Pre-assignment Details: A total of 799 participants were randomised in this study. Of these, a total of 797 participants were enrolled and received at least one dose of any study drug and represented the Safety population during the Double-Blind Treatment Phase (Parts 1 and 2 of the study). From the Double-Blind Treatment Phase, a total of 154 participants (at 53 sites) were enrolled into Open-Label Extension (OLE) Phase (Part 3 of the study).
Period: Double-Blind Treatment Phase
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Started | 266 | 271 | 260 | 0 | 0
Completed | 187 | 185 | 180 | 0 | 0
Not Completed | 79 | 86 | 80 | 0 | 0
Not completed — Death | 3 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 6 | 5 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 5 | 3 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0
Not completed — Participant/legal guardian decision | 7 | 8 | 8 | 0 | 0
Not completed — Parts 1 and 2 Termination by Sponsor | 62 | 68 | 63 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0
Period: Open-Label Extension (OLE) Phase
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Started | 0 | 0 | 0 | 49 | 105
Completed | 0 | 0 | 0 | 33 | 71
Not Completed | 0 | 0 | 0 | 16 | 34
Not completed — Death | 0 | 0 | 0 | 1 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 6
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 7
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6 | 15
Not completed — Other | 0 | 0 | 0 | 5 | 3

BASELINE CHARACTERISTICS:
Population: A total of 797 participants were enrolled into the Double-Blind Treatment phase of this study and the entire study. A subset (154) of these participants moved into the OLE phase of this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE]) | Total
Number analyzed (Participants) | 266 | 271 | 260 | 49 | 105 | 951
Age, Continuous [Mean (Standard Deviation); unit: years] — Parts 1 and 2 of the study. Population: Participants in the Double-Blind Treatment Phase of this study.
  years
    number analyzed (Participants) | 266 | 271 | 260 | 0 | 0 | 797
    (all) | 69.5 (7.5) | 70.3 (7.0) | 71.3 (7.1) |  |  | 70.4 (7.2)
Age, Continuous [Mean (Standard Deviation); unit: years] — Part 3 of the study. Population: Participants in the OLE Phase of this study.
  years
    number analyzed (Participants) | 0 | 0 | 0 | 49 | 105 | 154
    (all) |  |  |  | 75.5 (5.8) | 73.7 (7.3) | 74.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Parts 1 and 2 of the study. Population: Participants in the Double-Blind Treatment Phase of this study.
  Participants
    number analyzed (Participants) | 266 | 271 | 260 | 0 | 0 | 797
    Female | 149 | 152 | 152 | 0 | 0 | 453
    Male | 117 | 119 | 108 | 0 | 0 | 344
Sex: Female, Male [Count of Participants; unit: Participants] — Part 3 of the study. Population: Participants in the OLE Phase of this study.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 49 | 105 | 154
    Female | 0 | 0 | 0 | 27 | 64 | 91
    Male | 0 | 0 | 0 | 22 | 41 | 63
Race/Ethnicity, Customized [Number; unit: Participants] — Parts 1 and 2 of the study. Population: Participants in the Double-Blind Treatment Phase of this study.
  Participants
    Non-Hispanic: number analyzed (Participants) | 266 | 271 | 260 | 0 | 0 | 797
    Non-Hispanic | 217 | 221 | 210 |  |  | 648
    Hispanic: number analyzed (Participants) | 266 | 271 | 260 | 0 | 0 | 797
    Hispanic | 41 | 39 | 47 |  |  | 127
    American Indian or Alaska native: number analyzed (Participants) | 266 | 271 | 260 | 0 | 0 | 797
    American Indian or Alaska native | 1 | 6 | 5 |  |  | 12
    Asian: number analyzed (Participants) | 266 | 271 | 260 | 0 | 0 | 797
    Asian | 9 | 4 | 7 |  |  | 20
    Black: number analyzed (Participants) | 266 | 271 | 260 | 0 | 0 | 797
    Black | 1 | 2 | 2 |  |  | 5
    White: number analyzed (Participants) | 266 | 271 | 260 | 0 | 0 | 797
    White | 239 | 252 | 239 |  |  | 730
    Not Available: number analyzed (Participants) | 266 | 271 | 260 | 0 | 0 | 797
    Not Available | 24 | 18 | 10 |  |  | 52
Race/Ethnicity, Customized [Number; unit: Participants] — Part 3 of the study. Population: Participants in the OLE Phase of this study.
  Participants
    Non-Hispanic: number analyzed (Participants) | 0 | 0 | 0 | 49 | 105 | 154
    Non-Hispanic |  |  |  | 39 | 88 | 127
    Hispanic: number analyzed (Participants) | 0 | 0 | 0 | 49 | 105 | 154
    Hispanic |  |  |  | 10 | 17 | 27
    American Indian or Alaska native: number analyzed (Participants) | 0 | 0 | 0 | 49 | 105 | 154
    American Indian or Alaska native |  |  |  | 0 | 3 | 3
    Asian: number analyzed (Participants) | 0 | 0 | 0 | 49 | 105 | 154
    Asian |  |  |  | 2 | 0 | 2
    White: number analyzed (Participants) | 0 | 0 | 0 | 49 | 105 | 154
    White |  |  |  | 42 | 101 | 143
    Unknown: number analyzed (Participants) | 0 | 0 | 0 | 49 | 105 | 154
    Unknown |  |  |  | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB) Total Score at Week 104 (Double-Blind Treatment Phase)
Description: The CDR (Clinical Dementia Rating) is obtained through semi-structured interviews of participants and informants, and cognitive functioning is rated in six domains of functioning: memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care. Each domain is rated on a five-point scale of functioning as follows: 0, no impairment; 0.5, questionable impairment; 1, mild impairment; 2, moderate impairment; and 3, severe impairment. The CDR-SOB (Clinical Dementia Rating-Sum of Boxes) is based on summing each of the domain box scores with total scores ranging from 0-18, where lower total scores represent better outcomes and higher total scores represent worse outcomes.
Time Frame: Baseline, Week 104
Population: The Intent-To-Treat (ITT) population was defined as all participants who had received any dose of study treatment and had at least one post-baseline assessment of CDR-SOB. Data presented below is only for participants included in the actual analysis.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 104 | 105 | 100
Scores on a Scale | 1.19 (1.68) | 1.41 (2.02) | 1.47 (1.89)
Statistical Analysis 1: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 105 mg (Parts 1 and 2); Test type: Superiority; p = 0.6744, Mixed Models Analysis; Effect Size = -0.044, 95% CI 2-sided [-0.248 to 0.161]
Statistical Analysis 2: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 225 mg (Parts 1 and 2); Test type: Superiority; p = 0.4494, Mixed Models Analysis; Effect Size = -0.085, 95% CI 2-sided [-0.304 to 0.135]

2. Primary Outcome: Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) (OLE Phase)
Description: An Adverse Event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up until a maximum of 5 years
Population: The Safety population was defined as all participants who had received at least one dose of Gantenerumab during the OLE phase. All participants in the Safety population also had at least one post-OLE baseline MRI.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 49 | 105
Participants
  AEs | 46 | 100
  SAEs | 18 | 28

3. Secondary Outcome: Mean Change From Baseline in Alzheimer Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog-11) Scores at Week 104 (Double-Blind Treatment Phase)
Description: The ADAS-Cog-11 assesses multiple cognitive domains including memory, comprehension, praxis, orientation, and spontaneous speech. Most of these are assessed by tests although some are rated by the clinician on a 5-point scale. The score range for ADAS-Cog-11 is from 0 to 70 with higher scores representing severe dysfunction.
Time Frame: Baseline, Week 104
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 105 | 104 | 100
Scores on a Scale | 3.68 (6.64) | 3.52 (6.28) | 3.97 (6.89)
Statistical Analysis 1: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 105 mg (Parts 1 and 2); Test type: Superiority; p = 0.7458, Mixed Models Analysis; Effect Size = 0.035, 95% CI 2-sided [-0.179 to 0.250]
Statistical Analysis 2: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 225 mg (Parts 1 and 2); Test type: Superiority; p = 0.723, Mixed Models Analysis; Effect Size = 0.042, 95% CI 2-sided [-0.191 to 0.275]

4. Secondary Outcome: Time to Onset of Dementia at Week 104 (Double-Blind Treatment Phase)
Description: Time to Onset of Dementia was defined as the time interval between the first treatment date and the date that participant is assessed as having Alzheimer-type dementia by investigators.
Time Frame: Baseline, Week 104
Population: The Intent-To-Treat (ITT) population was defined as all participants who had received any dose of study treatment and had at least one post-baseline assessment of CDR-SOB.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 91 | 95 | 91
Days | 63.64 [56.63 to 69.82] | 62.98 [56.00 to 69.16] | 70.64 [63.34 to 76.75]

5. Secondary Outcome: Mean Change From Baseline in Cambridge Neuropsychological Test Automated Battery (CANTAB) Composite Score at Week 104 (Double-Blind Treatment Phase)
Description: The Cambridge Neuropsychological Test Automated Battery (CANTAB) ® is a cognitive test battery that incorporates a variety of executive and memory tasks in order to assess neuropsychological function. The end outcome as reported below, is a Z-Composite Score. The score range of the Z-Composite Score is from (-) infinity to (+) infinity with a score of zero representing the population mean, lower (negative) scores representing poorer cognitive outcomes and higher (positive) scores representing better cognitive outcomes.
Time Frame: Baseline, Week 104
Population: The Intent-To-Treat (ITT) population was defined as all participants who had received any dose of study treatment and had at least one post-baseline assessment of CDR-SOB. The Placebo Match Gantenerumab 225mg (Parts 1 and 2) arm consisted of participants with the ApoE 2e4 mutation who were excluded from the Gantenerumab 225 mg (Parts 1 and 2) arm. Data presented below is only for participants included in the actual analysis.
Measure: Mean (Standard Deviation); unit: Z-Score
Groups:
- Placebo Match Gantenerumab 225 mg (Parts 1 and 2): Participants with Alzheimer's disease received matching Placebo to Gantenerumab 225 mg by SC injection q4w for 104 weeks or approximately 2 years during Part 1 of the study. Participants who completed the Week 104 visit were given an option to continue the treatment received during Part 1, for 2 additional years in Part 2.
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo Match Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 90 | 87 | 80 | 73
Z-Score | -1.72 (2.99) | -1.37 (2.74) | -1.4 (3.11) | -1.93 (3.08)

6. Secondary Outcome: Mean Change From Baseline in Free and Cued Selective Reminding Test (FCSRT) Score at Week 104 (Double-Blind Treatment Phase)
Description: FCSRT assesses verbal episodic memory. Performances in free recalls, cued recalls and in a recognition task were analyzed, as the process of encoding is controlled. Participants were asked to remember a list of 16 words. Three tasks of free and cued recalls, as well as 1 recognition task and one delayed recall give the scores. Total recall was obtained by the addition of cued recalls to free recalls. Maximum score is 48 for immediate: 16 words multiplied by (*) 3 corresponding to immediate free recall + immediate cued recall + immediate recognition test. Maximum score is 64 (better score) when delayed recall: 16 words*4. The minimum score is 0 (worse).
Time Frame: Baseline, Week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo Match Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 100 | 102 | 97 | 79
Scores on a Scale | -4.05 (8.73) | -4.11 (8.57) | -6.42 (8.45) | -4.05 (8.68)

7. Secondary Outcome: Mean Change From Baseline in Functional Activities Questionnaire (FAQ) Score at Week 104 (Double-Blind Treatment Phase)
Description: Participants completed the FAQ for physical function. Overall scores ranged from 0 (independent) to 30 (dependent) where lower scores represented an improvement in physical function.
Time Frame: Baseline, Week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Groups:
- Placebo (Parts 1 and 2): Participants with Alzheimer's disease received Placebo SC injection (Q4W) for 104 weeks or approximately 2 years during Part 1 of the study. Participants who completed the Week 104 visit were given an option to continue the treatment received during Part 1, for 2 additional years in Part 2.
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo Match Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 105 | 104 | 99 | 84
Scores on a Scale | 3.59 (4.93) | 4.89 (6.2) | 4.03 (5.75) | 3.6 (4.93)
Statistical Analysis 1: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 105 mg (Parts 1 and 2); Test type: Superiority; p = 0.0825, Mixed Models Analysis; Effect Size = -0.191, 95% CI 2-sided [-0.407 to 0.025]
Statistical Analysis 2: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 225 mg (Parts 1 and 2); Test type: Superiority; p = 0.7171, Mixed Models Analysis; Effect Size = 0.043, 95% CI 2-sided [-0.19 to 0.276]

8. Secondary Outcome: Mean Change From Baseline in CDR-Global Score at Week 104 (Double-Blind Treatment Phase)
Description: The CDR-GS represents a semi-structured interview which rates impairment in 6 categories (memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care) on a 5-point scale in which CDR 0 = no dementia and CDR 0.5, 1, 2 or 3 = questionable, mild, moderate or severe dementia respectively. The range in scores for the CDR-GS is from 0 to 3 and a high score on the CDR-GS would indicate a high disease severity.
Time Frame: Baseline, Week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo Match Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 104 | 105 | 100 | 83
Scores on a Scale | 0.1 (0.29) | 0.18 (0.36) | 0.14 (0.33) | 0.1 (0.31)

9. Secondary Outcome: Mean Change From Baseline in Neuropsychiatric Inventory (NPI) Questionnaire Score at Week 104 (Double-Blind Treatment Phase)
Description: The NPI is a retrospective (to 1 month) caregiver-informant interview assessing frequency and severity of 12 neuropsychiatric symptom domains. The NPI score is based on the sum of the severity ratings (0=absent, 1=mild, 3=severe). The 12 symptom domains include delusions, hallucinations, agitation/aggression, dysphoria/depression, anxiety, euphoria/elation, apathy/indifference, disinhibition, irritability/lability, aberrant motor behaviors, nighttime behavioral disturbances, and appetite/eating abnormalities. The NPI severity score is based on severity ratings (0=absent, 1=mild to 3=severe).
Time Frame: Baseline, Week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo Match Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 103 | 105 | 99 | 82
Scores on a Scale | 0.6 (3.22) | 0.39 (2.57) | 0.34 (2.84) | 0.72 (3.35)

10. Secondary Outcome: Percentage Change From Baseline in Cerebrospinal Fluid Biomarkers (Phosphorylated-tau [P-tau], Amyloid Beta 1-42 [Abeta 1-42], Total Tau [T-tau]) at Week 104 (Double-Blind Treatment Phase)
Description: CSF biomarker phospho-tau (p-tau) is an indicator of neuronal injury and neurodegeneration. An elevation in levels of tau, as well as specific p-tau species, is thought to be a marker for progressive cellular degeneration in AD.
Time Frame: Baseline, Week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo Match Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 72 | 71 | 66 | 56
Percentage Change
  p-tau (Week 104) | 2.77 (20.69) | -4.78 (11.9) | -7.34 (10.09) | 2.84 (23.19)
  t-tau (Week 104) | 3.43 (19.95) | -1.36 (12.89) | -2.12 (11.01) | 3.46 (22.32)
  Abeta (Week 104): number analyzed (Participants) | 69 | 64 | 65 | 56
  Abeta (Week 104) | 4.87 (36.14) | 2.45 (24.57) | 15.2 (45.24) | 4.3 (39.31)
Statistical Analysis 1: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 105 mg (Parts 1 and 2); Statistical analysis of the Abeta 1-42 CSF biomarker between "Placebo (Parts 1 and 2)" and "Gantenerumab 105 mg (Parts 1 and 2)" treatment arms at Week 104; Test type: Superiority; p = 0.9734, Mixed Models Analysis
Statistical Analysis 2: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 225 mg (Parts 1 and 2); Statistical analysis of the Abeta 1-42 CSF biomarker between "Placebo (Parts 1 and 2)" and "Gantenerumab 225 mg (Parts 1 and 2)" treatment arms at Week 104; Test type: Superiority; p = 0.0629, Mixed Models Analysis
Statistical Analysis 3: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 105 mg (Parts 1 and 2); Statistical analysis of the p-tau CSF biomarker between "Placebo (Parts 1 and 2)" and "Gantenerumab 105 mg (Parts 1 and 2)" treatment arms at Week 104; Test type: Superiority; p = 0.0084, Mixed Models Analysis
Statistical Analysis 4: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 225 mg (Parts 1 and 2); Statistical analysis of the p-tau CSF biomarker between "Placebo (Parts 1 and 2)" and "Gantenerumab 225 mg (Parts 1 and 2)" treatment arms at Week 104; Test type: Superiority; p = 0.0003, Mixed Models Analysis
Statistical Analysis 5: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 105 mg (Parts 1 and 2); Statistical analysis of the t-tau CSF biomarker between "Placebo (Parts 1 and 2)" and "Gantenerumab 105 mg (Parts 1 and 2)" treatment arms at Week 104; Test type: Superiority; p = 0.0903, Mixed Models Analysis
Statistical Analysis 6: Comparison: Placebo (Parts 1 and 2) vs Gantenerumab 225 mg (Parts 1 and 2); Statistical analysis of the t-tau CSF biomarker between "Placebo (Parts 1 and 2)" and "Gantenerumab 225 mg (Parts 1 and 2)" treatment arms at Week 104; Test type: Superiority; p = 0.0434, Mixed Models Analysis

11. Secondary Outcome: Percentage Change From Baseline in Hippocampal Volume at Week 104 (Double-Blind Treatment Phase)
Description: Change from baseline in hippocampal right volume (HRV) and hippocampal left volume (HLV) were analysed at Week 104 using magnetic resonance imaging.
Time Frame: Baseline, Week 104
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo Match Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 131 | 124 | 119 | 107
Percentage Change
  HRV (Week 104) | -7.61 (4.03) | -7.52 (3.96) | -7.34 (3.84) | -7.7 (4.01)
  HLV (Week 104) | -7.8 (4.28) | -7.76 (3.74) | -7.27 (3.78) | -8.12 (4.19)

12. Secondary Outcome: Percentage Change From Baseline in Cortical Composite Sustained Uptake Volume Ratio (SUVr) in Different Brain Regions at Week 156 (Double-Blind Treatment Phase)
Description: The different regions of the brain that were analyzed included cerebellum gray, whole cerebellum, composite white matter, subcortical white matter, pons and composite reference.
Time Frame: Baseline, Week 156
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo Match Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 6 | 4 | 10 | 4
Percentage Change
  Cerebellum gray (Week 156) | 6.26 (9.1) | 2.7 (10.59) | -8.36 (9.11) | 5.95 (11.13)
  Whole Cerebellum (Week 156) | 5.41 (7.13) | 2.07 (8.65) | -8.44 (8.06) | 5.17 (8.66)
  Composite White Matter (Week 156) | 2.75 (3.18) | -0.87 (2.95) | -4.86 (6.35) | 3.07 (2.07)
  Subcortical White Matter (Week 156) | 4.83 (4.95) | 1.69 (4.45) | -0.42 (8.26) | 4.59 (0.55)
  Pons (Week 156) | 1.72 (2.51) | -2.83 (3.39) | -6.99 (5.65) | 2.1 (2.73)
  Composite Reference (Week 156) | 4.5 (3.48) | 1.19 (5.63) | -6.75 (6.1) | 4.46 (4.49)

13. Secondary Outcome: Gantenerumab Plasma Concentrations at Different Time Points (Double-Blind Treatment Phase)
Description: The PK analyses includes tabulation of plasma concentration data and summarisation of plasma concentrations by visits with participants grouped according to treatment received. Descriptive summary statistics for the Arithmetic Mean and Standard Deviation are presented below.
Time Frame: Pre-Dose: Weeks 8, 20, 44, 68 and 100; Post-Dose: Weeks 1, 53 and 101
Population: The Intent-To-Treat (ITT) population was defined as all participants who had received any dose of study treatment and had at least one post-baseline assessment of CDR-SOB. Data presented below is only for participants included in the actual analysis and note that participants who received dose reduction were excluded from this PK analysis.
Measure: Mean (Standard Deviation); unit: µg/ml (micrograms per milliliter)
Arm/Group | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 239 | 227
µg/ml (micrograms per milliliter)
  Week 1 (Post-Dose) | 3.56 (2.36) | 7.4 (4.28)
  Week 8 (Pre-Dose): number analyzed (Participants) | 237 | 225
  Week 8 (Pre-Dose) | 2.87 (1.84) | 5.92 (3.16)
  Week 20 (Pre-Dose): number analyzed (Participants) | 228 | 220
  Week 20 (Pre-Dose) | 3.7 (2.15) | 7.66 (4.14)
  Week 44 (Pre-Dose): number analyzed (Participants) | 212 | 199
  Week 44 (Pre-Dose) | 4.08 (2.44) | 8.22 (4.51)
  Week 53 (Post-Dose): number analyzed (Participants) | 195 | 185
  Week 53 (Post-Dose) | 6.77 (3.94) | 15 (9.34)
  Week 68 (Pre-Dose): number analyzed (Participants) | 165 | 155
  Week 68 (Pre-Dose) | 3.95 (2.35) | 8.91 (4.86)
  Week 100 (Pre-Dose): number analyzed (Participants) | 98 | 86
  Week 100 (Pre-Dose) | 4.35 (2.34) | 9.4 (4.69)
  Week 101 (Post-Dose): number analyzed (Participants) | 95 | 77
  Week 101 (Post-Dose) | 7.32 (3.53) | 16.63 (7.96)

14. Secondary Outcome: Mean Change From Baseline in Mini Mental State Exam (MMSE) Score at Week 104 (Double-Blind Treatment Phase)
Description: The MMSE is a brief, practical screening test for cognitive dysfunction. The test consists of five sections (orientation, registration, attention-calculation, recall, and language); the total score can range from 0 to 30, with a higher score indicating better function. A positive change score indicates improvement.
Time Frame: Baseline, Week 104
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 104 | 105 | 99
Scores on a Scale | -2.31 (3.23) | -2.46 (3.68) | -2.25 (3.31)

15. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Serious Adverse Events (SAEs) (Double-Blind Treatment Phase)
Description: as for outcome 2
Time Frame: Baseline up until a maximum of 4.5 years
Population: The Safety population was defined as all participants who had received at least one dose of study drug, regardless of whether the participant withdrew prematurely or not. All safety data was analyzed according to study drug actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 266 | 271 | 260
Participants
  AEs | 250 | 241 | 240
  SAEs | 55 | 48 | 46

16. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) (Double-Blind Treatment Phase)
Description: Participants were considered positive or negative for ADA based on their baseline and post-baseline sample results. The number and percentage of participants with confirmed positive ADA levels were determined for Gantenerumab and Placebo groups. The prevalence of ADA at baseline was calculated as the proportion of participants with confirmed positive ADA levels at baseline relative to the total number of participants with a sample available at baseline. The incidence of treatment-emergent ADAs was determined as the proportion of participants with confirmed post-baseline positive ADAs relative to the total number of participants that had at least one post-baseline sample available for ADA analysis.
Time Frame: Baseline up until a maximum of 4.5 years
Population: The Safety population was defined as all participants who had received at least one dose of study drug, regardless of whether the participant withdrew prematurely or not. All safety data was analyzed according to study drug actually received. Data presented below is only for participants included in the actual analysis.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2)
Number analyzed (Participants) | 259 | 266 | 256
Percentage of Participants
  Baseline ADAs | 5.8 | 7.5 | 5.5
  Treatment Emergent ADAs: number analyzed (Participants) | 259 | 258 | 250
  Treatment Emergent ADAs | 5.0 | 7.0 | 6.4

17. Secondary Outcome: Mean Change From Baseline in Alzheimer Disease Assessment Scale-Cognitive Subscale 11 (ADAS-Cog-11) Scores at Week 156 (OLE Phase)
Description: as for outcome 3
Time Frame: Baseline, Week 156
Population: The Safety population was defined as all participants who had received at least one dose of Gantenerumab during the OLE phase. All participants in the Safety population also had at least one post-OLE baseline MRI. Data presented below is only for participants included in the actual analysis.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 21 | 51
Scores on a Scale | 5.8 (7.3) | 8.9 (9.7)

18. Secondary Outcome: Mean Change From Baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SOB) Total Score at Week 156 (OLE Phase)
Description: as for outcome 1
Time Frame: Baseline, Week 156
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 21 | 52
Scores on a Scale | 3.3 (2.4) | 2.8 (3.0)

19. Secondary Outcome: Mean Change From Baseline in Alzheimer Disease Assessment Scale-Cognitive Subscale 13 (ADAS-Cog-13) Scores at Week 156 (OLE Phase)
Description: The ADAS-Cog-13 assesses multiple cognitive domains including memory, comprehension, praxis, orientation, and spontaneous speech. The score range for ADAS-Cog-13 is from 0 to 85 with higher scores representing severe dysfunction.
Time Frame: Baseline, Week 156
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 21 | 51
Scores on a Scale | 8.0 (8.2) | 10.4 (10.6)

20. Secondary Outcome: Time to Onset of Dementia at Week 156 (OLE Phase)
Description: as for outcome 4
Time Frame: Baseline, Week 156
Population: as for outcome 17
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 3 | 14
Days | 38.18 [9.90 to 66.97] | 50.82 [32.04 to 66.87]

21. Secondary Outcome: Mean Change From Baseline in Free and Cued Selective Reminding Test (FCSRT) Score at Week 156 (OLE Phase)
Description: as for outcome 6
Time Frame: Baseline, Week 156
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 22 | 51
Scores on a Scale | -7.7 (9.3) | -4.1 (8.3)

22. Secondary Outcome: Mean Change From Baseline in Functional Activities Questionnaire (FAQ) Score at Week 156 (OLE Phase)
Description: as for outcome 7
Time Frame: Baseline, Week 156
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 22 | 52
Scores on a Scale | 8.1 (5.3) | 6.8 (6.8)

23. Secondary Outcome: Mean Change From Baseline in CDR-Global Score at Week 156 (OLE Phase)
Description: as for outcome 8
Time Frame: Baseline, Week 156
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 21 | 52
Scores on a Scale | 0.6 (0.6) | 0.5 (0.6)

24. Secondary Outcome: Percentage Change From Baseline in Hippocampal Volume at Week 152 (OLE Phase)
Description: Change from baseline in hippocampal right volume (HRV) and hippocampal left volume (HLV) were analysed at Week 152 using magnetic resonance imaging.
Time Frame: Baseline, Week 152
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 18 | 51
Percentage Change
  HRV (Week 152) | 16.7 (8.4) | 16.1 (8.2)
  HLV (Week 152) | 16.2 (13.0) | 18.0 (8.9)

25. Secondary Outcome: Percentage Change From Baseline in Cortical Composite Sustained Uptake Volume Ratio (SUVr) in Different Brain Regions at Week 156 (OLE Phase)
Description: The regions of the brain that were analyzed included cerebellum gray and composite reference.
Time Frame: Baseline, Week 156
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 2
Percentage Change
  Cerebellum gray (Week 156) | -0.2 (0.2)
  Composite Reference (Week 156) | -41.4 (29.9)

26. Secondary Outcome: Gantenerumab Plasma Concentrations at Different Time Points (OLE Phase)
Description: as for outcome 13
Time Frame: Pre-Dose: Weeks 64, 100, 104, 136, 156 and 208; Post-Dose: Week 101
Population: The Safety population was defined as all participants who had received at least one dose of Gantenerumab during the OLE phase. All participants in the Safety population also had at least one post-OLE baseline MRI. Data presented below is only for participants included in the actual analysis and note that participants who received dose reduction were excluded from this PK analysis.
Measure: Mean (Standard Deviation); unit: µg/ml (micrograms per milliliter)
Groups:
- Gantenerumab 1200 mg (Part 3 Open-Label Extension [OLE]): Participants with Alzheimer's disease who had received Gantenerumab by SC injection in Part 1 or Part 2, now received Gantenerumab at a dose of 1200 mg by SC injection every 4 weeks (Q4W) for up to 5 additional years.
Arm/Group | Gantenerumab 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 99
µg/ml (micrograms per milliliter)
  Week 64 (Pre-Dose) | 33.0 (21.7)
  Week 100 (Pre-Dose): number analyzed (Participants) | 89
  Week 100 (Pre-Dose) | 39.2 (22.7)
  Week 101 (Post-Dose): number analyzed (Participants) | 88
  Week 101 (Post-Dose) | 80.5 (37.8)
  Week 104 (Pre-Dose): number analyzed (Participants) | 91
  Week 104 (Pre-Dose) | 40.5 (22.5)
  Week 136 (Pre-Dose): number analyzed (Participants) | 83
  Week 136 (Pre-Dose) | 45.2 (22.4)
  Week 156 (Pre-Dose): number analyzed (Participants) | 93
  Week 156 (Pre-Dose) | 39.6 (28.2)
  Week 208 (Pre-Dose): number analyzed (Participants) | 26
  Week 208 (Pre-Dose) | 37.1 (29.2)

27. Secondary Outcome: Mean Change From Baseline in Mini Mental State Exam (MMSE) Score at Week 156 (OLE Phase)
Description: as for outcome 14
Time Frame: Baseline, Week 156
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 22 | 53
Scores on a Scale | -4.3 (4.3) | -4.7 (4.6)

28. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADAs) (OLE Phase)
Description: Participants were considered positive or negative for ADA based on their baseline and post-baseline sample results. The number and percentage of participants with confirmed positive ADA levels were determined. The prevalence of ADA at baseline was calculated as the proportion of participants with confirmed positive ADA levels at baseline relative to the total number of participants with a sample available at baseline. The incidence of treatment-emergent ADAs was determined as the proportion of participants with confirmed post-baseline positive ADAs relative to the total number of participants that had at least one post-baseline sample available for ADA analysis.
Time Frame: Baseline up until a maximum of 5 years
Population: as for outcome 17
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
Number analyzed (Participants) | 49 | 104
Percentage of Participants
  Baseline ADAs | 2.0 | 5.8
  Treatment Emergent ADAs: number analyzed (Participants) | 46 | 102
  Treatment Emergent ADAs | 2.2 | 2.9

ADVERSE EVENTS:
Time Frame: Baseline up until a maximum of 9.5 years
Arm/Group | Placebo (Parts 1 and 2) | Gantenerumab 105 mg (Parts 1 and 2) | Gantenerumab 225 mg (Parts 1 and 2) | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE])
All-Cause Mortality (participants affected / at risk) | 6/266 | 0/271 | 2/260 | 1/49 | 3/105
Serious Adverse Events (participants affected / at risk) | 55/266 | 48/271 | 46/260 | 18/49 | 28/105
Other Adverse Events (participants affected / at risk) | 163/266 | 188/271 | 189/260 | 40/49 | 87/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Parts 1 and 2) (N=266) | Gantenerumab 105 mg (Parts 1 and 2) (N=271) | Gantenerumab 225 mg (Parts 1 and 2) (N=260) | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) (N=49) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE]) (N=105)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARIA-E (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dementia with Lewy bodies (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retrograde amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Delirium (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropsychiatric symptoms (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal behaviour (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rotator cuff repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urethral caruncle removal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Myocardial rupture (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus arrest (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes insipidus (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type I hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radial nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bone sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation mucositis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Behavioral and psychological symptoms of dementia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral dilation procedure (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (Parts 1 and 2) (N=266) | Gantenerumab 105 mg (Parts 1 and 2) (N=271) | Gantenerumab 225 mg (Parts 1 and 2) (N=260) | Placebo (Parts 1 and 2) Switched to Gantenerumab Up to 1200mg (Part 3 Open-Label Extension [OLE]) (N=49) | Gantenerumab Up to 1200 mg (Part 3 Open-Label Extension [OLE]) (N=105)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 13 (18) | 15 (22) | 15 (18) | 3 (3) | 11 (14)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (9)
Injection site erythema (General disorders) | 3 (3) | 29 (133) | 35 (114) | 17 (196) | 36 (359)
Bronchitis (Infections and infestations) | 10 (10) | 10 (12) | 14 (18) | 3 (3) | 7 (9)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Influenza (Infections and infestations) | 13 (14) | 13 (18) | 15 (17) | 3 (4) | 7 (8)
Nasopharyngitis (Infections and infestations) | 17 (34) | 30 (40) | 20 (35) | 7 (7) | 15 (23)
Upper respiratory tract infection (Infections and infestations) | 11 (14) | 13 (15) | 18 (21) | 5 (5) | 10 (19)
Urinary tract infection (Infections and infestations) | 25 (37) | 16 (25) | 22 (38) | 4 (6) | 15 (25)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 5 (5)
Fall (Injury, poisoning and procedural complications) | 28 (42) | 23 (32) | 27 (38) | 13 (20) | 17 (29)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (29) | 12 (14) | 16 (17) | 2 (2) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (33) | 16 (18) | 26 (32) | 2 (2) | 10 (10)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 31 (51) | 58 (92) | 36 (64) | 7 (12) | 17 (44)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 2 (2) | 18 (20) | 34 (36) | 12 (21) | 29 (45)
Dizziness (Nervous system disorders) | 21 (21) | 21 (27) | 26 (35) | 4 (5) | 14 (18)
Headache (Nervous system disorders) | 36 (50) | 34 (47) | 25 (36) | 7 (11) | 12 (18)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 8 (10)
Anxiety (Psychiatric disorders) | 18 (23) | 20 (20) | 16 (16) | 2 (2) | 7 (8)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 8 (8)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 6 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 11 (13) | 13 (13) | 5 (5) | 8 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 18 (20) | 11 (11) | 20 (23) | 2 (2) | 8 (11)
Depression (Psychiatric disorders) | 13 (14) | 23 (23) | 25 (25) | 0 (0) | 0 (0)
Fatigue (General disorders) | 8 (8) | 7 (7) | 15 (20) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 6 (7) | 5 (5) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-07-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT01224106/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/06/NCT01224106/SAP_001.pdf